CLINICAL TRIAL: NCT06860451
Title: To Explore the Neural Processing Mechanism of Cerebellum Involved in Facial Expression Recognition Based on Transcranial Magnetic Stimulation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Liqing Yao, Director, Department of Rehabilitation Medicine, the Second Affiliated Hospital of Kunming Medical University, The Second Affiliated Hospital of Kunming Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Shen-PJ-Ke-2024-201
Record Dates: First submitted 2024-11-14; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Post-stroke Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Right cerebellar intervention group (Experimental): The single-pulse TMS intervention in right cerebellum
  Interventions: Device: TMS
- Left cerebellar intervention group (Experimental): The single-pulse TMS intervention in left cerebellum
  Interventions: Device: TMS
- The vermis cerebellar intervention group (Experimental): The single-pulse TMS intervention in vermis cerebellar
  Interventions: Device: TMS
- Sham TMS (Sham Comparator): The TMS coil was placed at the cerebellar site but tilted 90° to prevent effective magnetic field penetration.
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — The single-pulse TMS

SUMMARY:
Experiment 1: Utilizing a transcranial magnetic stimulation-electroencephalography/functional near-infrared spectroscopy system, the investigators aim to determine whether transcranial magnetic stimulation of the cerebellum can alter neural oscillations and blood flow changes in the prefrontal cortex. The investigators will recruit 80 healthy volunteers and 80 stroke patients with middle cerebral artery infarction, each meeting the inclusion criteria. Twenty healthy volunteers and twenty patients will be randomly selected to receive a single-pulse transcranial magnetic stimulation (TMS) to the cerebellar vermis. The investigators will record cerebellar transcranial evoked potentials (TEP) in the EEG to assess cerebellar cortical excitability and inhibition and evaluate individuals using functional near-infrared spectroscopy to analyze changes in prefrontal blood flow and brain networks. The other 40 healthy volunteers and 40 patients will receive a single-pulse TMS to the right or left cerebellum, and similar assessments will be made. The remaining 20 healthy volunteers and 20 patients will receive a sham iTBS, with similar assessments.

Experiment 2: Through a facial expression recognition task, this experiment aims to clarify the cerebellum's increased perception of negative emotions, thereby achieving a rebalance from "controlled" to "automatic" regulation of negative emotions, ultimately playing a role in "automatic" emotional adjustment. The 80 healthy volunteers from Experiment 1 will be equally divided into four groups based on stimulation site: the cerebellar vermis; the right cerebellum; the left cerebellum; the sham stimulation. Each group will perform the facial expression recognition task during the TMS stimulation. The investigators will collect functional near-infrared spectroscopy and task-based EEG data from the participants during stimulation while also recording their response times, accuracy rates, and completion conditions, including their tolerance of the experiment and any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Onset of stroke <6 months ago, or >6 months since the last stroke event;
* Age >=18 years and <85 years (as the probability of Vascular Cognitive Impairment increases above 85);
* Patients with damage in the middle cerebral artery territory;
* NIHSS >4 and <26;
* mRS score >=2;
* Completion of CT or MRI;
* No neurological or psychiatric disorders; no impairment of consciousness; able to comply with relevant treatments; no severe cognitive dysfunction (MMSE >=15);
* All participants are right-handed; Sign the informed consent form.

Exclusion Criteria:

* History of epilepsy or psychiatric disorders (including depression, anxiety, or schizophrenia);
* Severe comorbidities;
* History of medication use: benzodiazepines, baclofen, antidepressants;
* Non-compliance with the treatment plan;
* Acute-phase cerebral hemorrhage, acute infectious diseases;
* Severe suicidal tendencies in individuals with depression;
* Individuals suffering from severe headaches, high blood pressure, malignant tumors, open wounds, vascular embolism, leukopenia, etc.;
* Severe alcohol abuse;
* History of cranial surgery, individuals with metal implants in the brain;
* Individuals with an implanted cardiac pacemaker;
* NIHSS >26, MMSE <15;
* Any disease likely to prevent the patient from surviving more than one month;
* Pregnant individuals.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-03-25 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Electroencephalogram | Day 1
  EEG power in the delta, theta, alpha, beta band: the power spectral density (PSD) in unit^2/Hz Functional connectivity---Phase locking value (PLV): The value of PLV ranges from 0 to 1 Event related potentials in amplitude/μV
Functional near - infrared spectroscopy , fNIRS | Day 1
  Hemodynamic curve (HbO) in μM

SECONDARY OUTCOMES:
Mini-mental state examination,MMSE | Day 1
  Mini-mental state examination,MMSE: A score of 27-30: normal; Score < 27: cognitive impairment.
Montreal Cognitive Assessment, MoCA | Day 1
  Montreal Cognitive Assessment, MoCA: The total score of the scale is 30 points, and the test result shows that the normal value is ≥26 points.
Hamilton Depression Scale，HAMD | Day 1
  Hamilton Depression Scale，HAMD: A total score of more than 35 May indicate severe depression.
Hamilton Anxiety Scale，HAMA | Day 1
  Hamilton Anxiety Scale，HAMA: The total score ≥29, may be severe anxiety; ≥21 points, there must be obvious anxiety; ≥14 points, definitely have anxiety; More than 7 points, may have anxiety; If the score is less than 7, there is no anxiety symptom
Montgomery-Asberg Depression Rating Scale，MADRS | Day 1
  Montgomery-Asberg Depression Rating Scale，MADRS: Extreme depression: MADRS >35; Major depression: MADRS >30; Moderate depression: MADRS >22; Mild depression: MADRS >12; Remission stage: MADRS <12.
Quick Inventory of Depressive Symptomatology Self-Report, QIDS-SR16 | Day 1
  Quick Inventory of Depressive Symptomatology Self-Report, QIDS-SR16: The total score is calculated on a scale of 0 to 27, with higher scores being associated with higher levels of depression.
Response time | Day 1
  Recording their response times in seconds: The average reaction time of subjects in the facial expression recognition task to judge each facial expression picture.
Accuracy rates | Day 1
  Recording their accuracy rates in % during the task: The average correct rate at which subjects judged each expression picture in the facial expression recognition task.

IPD SHARING:
Plan to Share IPD: No